CLINICAL TRIAL: NCT04959110
Title: Citrate Pharmacokinetics in Critically Ill Liver Failure Patients Receiving CRRT
Acronym: Citrate PK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Director of Excellence Center for Critical Care Nephrology, Chulalongkorn University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB.694/63
Record Dates: First submitted 2021-06-09; First posted 2021-07-13 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Citrate Toxicity; Regional Citrate Anticoagulation; Liver Failure, Acute; Liver Failure, Acute on Chronic; Pharmacokinetic; Continuous Renal Replacement Therapy
Keywords: Regional citrate anticoagulation; Liver failure; Pharmacokinetics; CRRT; Cirrhosis
MeSH Terms: conditions — Liver Failure, Acute; Acute-On-Chronic Liver Failure; Liver Failure; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Liver Failure (Experimental): Acute liver failure critically ill patients receiving CRRT
  Interventions: Diagnostic Test: Pharmacokinetic study
- Acute on top Chronic Liver Failure (Experimental): Acute on top chronic liver failure critically ill patients receiving CRRT
  Interventions: Diagnostic Test: Pharmacokinetic study

INTERVENTIONS:
Diagnostic Test: Pharmacokinetic study — * Start CVVH session with isotonic citrate solution (13.3 mmol/L) as predilution, targeting citrate dose at 3 mmol/L
  * Blood samples collection at pre-filter for citrate concentration, blood gas, electrolyte and ionized calcium and magnesium
  * In addition, 10 minutes after the end of citrate infusion, blood samples were taken simultaneously from both pre-filter and post-filter to calculate citrate clearance by filter

SUMMARY:
Citrate has been proposed as anticoagulation of choice in continuous renal replacement therapy (CRRT). However, little is known about the pharmacokinetics (PKs) and metabolism of citrate in liver failure patients who require CRRT with regional citrate anticoagulation (RCA).

DETAILED DESCRIPTION:
This study aimed to evaluate citrate PKs, metabolic complications, and clinical outcomes among critically ill acute liver failure (ALF) and acute on top chronic liver failure (ACLF) patients receiving CRRT.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill ALF or ACLF adult patients with AKI
* aged ≥ 18 y old
* Currently receiving CRRT.

Exclusion Criteria:

* severe acidosis (pH < 7.1) or severe alkalosis (pH > 7.55)
* blood transfusion within 24 h prior to the study
* use of citrate-containing medications
* severe hypocalcemia (serum ionized calcium < 0.8 mmol/L)
* use of heparin as anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Citrate clearance | 4 hours
  Citrate clearance by body

SECONDARY OUTCOMES:
Citrate accumulation | 4 hours
  Number of total calcium to ionized calcium ratio > 2.5 with acidosis with hypocalcemia
Tmax | 2 hours
  Time to maximum concentration of citrate at 2 hours
Area under the time curve | 4 hours
  Area under the plasma concentration-time curve of citrate
Change of systemic ionized calcium | 4 hours
  Change in systemic ionized calcium in arterial blood gas during study
Change of ionized magnesium | 4 hours
  Change in systemic ionized magnesium in arterial blood gas during study
Change of bicarbonate | 4 hours
  Change of bicarbonate in arterial blood gas during study
Ratio of total calcium to systemic ionized calcium | 4 hours
  Number of patients with total calcium to systemic ionized calcium > 2.5 with or without metabolic acidosis

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn university, Bangkok, Thailand